CLINICAL TRIAL: NCT02902198
Title: Taste Physiology in Obese Volunteers Before and After Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: fMRI Taste 2
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucose; Sodium Glutamate; Quinine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Placebo preoperative (Placebo Comparator): Single intragastric instillation of 200ml tap water via nasogastric tube
  Interventions: Dietary Supplement: Placebo
- Placebo postoperative (Placebo Comparator): Single intragastric instillation of 200ml tap water via nasogastric tube
  Interventions: Dietary Supplement: Placebo
- Glucose preoperative (Active Comparator): Single intragastric instillation of 200ml tap water with 25g glucose via nasogastric tube
  Interventions: Dietary Supplement: Glucose
- Glucose postoperative (Active Comparator): Single intragastric instillation of 200ml tap water with 25g glucose via nasogastric tube
  Interventions: Dietary Supplement: Glucose
- Monosodium glutamate preoperative (Active Comparator): Single intragastric instillation of 200ml tap water with 1g monosodium glutamate via nasogastric tube
  Interventions: Dietary Supplement: Monosodium glutamate
- Monosodium glutamate postoperative (Active Comparator): Single intragastric instillation of 200ml tap water with 1g monosodium glutamate via nasogastric tube
  Interventions: Dietary Supplement: Monosodium glutamate
- Quinine preoperative (Active Comparator): Single intragastric instillation of 200ml tap water with 17mg quinine via nasogastric tube
  Interventions: Dietary Supplement: Quinine
- Quinine postoperative (Active Comparator): Single intragastric instillation of 200ml tap water with 17mg quinine via nasogastric tube
  Interventions: Dietary Supplement: Quinine

INTERVENTIONS:
Dietary Supplement: Placebo — Tap water 200ml
  Arms: Placebo postoperative; Placebo preoperative
Dietary Supplement: Glucose — 25g Glucose in 200ml tap water
  Arms: Glucose postoperative; Glucose preoperative
Dietary Supplement: Monosodium glutamate — 1g monosodium glutamate in 200ml tap water
  Arms: Monosodium glutamate postoperative; Monosodium glutamate preoperative
Dietary Supplement: Quinine — 17mg quinine in 200ml tap water
  Arms: Quinine postoperative; Quinine preoperative

SUMMARY:
The objective is to investigate neuro-anatomical correlates of gastrointestinal taste stimulation by means of functional MRI before and after bariatric surgery. Intragastric administration of glucose, monosodium glutamate, chloroquine and placebo is followed by functional brain MRI in obese humans before and 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients (BMI min 35kg/m2) scheduled for bariatric surgery
* right handed

Exclusion Criteria:

* cardiovascular disease
* neurologic/psychiatric disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Effect of tastants on cerebral blood flow measured by functional brain MRI | changes from baseline to one hour after treatment

SECONDARY OUTCOMES:
Effect of tastants plasma glucagon-like peptide (GLP-1) concentrations | changes from baseline to one hour after treatment
Effect of tastants plasma ghrelin concentrations | changes from baseline to one hour after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Prof, Study Chair — University Basel
Locations (1):
- University Hopital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No